CLINICAL TRIAL: NCT04085276
Title: A Randomized, Double-Blind, Multicenter, Phase III Study of Toripalimab(JS001) in Combination With Nab-Paclitaxel Versus Placebo Plus Nab-Paclitaxel for Patients With Metastatic or Recurrent Triple-Negative Breast Cancer With or Without Systemic Treatment (TORCHLIGHT)
Brief Title: Toripalimab in Combination With Nab-Paclitaxel For Patients With Metastatic or Recurrent Triple-Negative Breast Cancer (TNBC) With or Without Systemic Treatment
Acronym: TORCHLIGHT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-026-III-TNBC
Record Dates: First submitted 2019-07-25; First posted 2019-09-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS001 Plus Nab-Paclitaxel (Experimental): Patients will receive both JS001 and Nab-Paclitaxel.
  Interventions: Drug: JS001; Drug: Nab-Paclitaxel
- Placebo Plus Nab-Paclitaxel (Placebo Comparator): Patients will receive both placebo and Nab-Paclitaxel.
  Interventions: Drug: Placebo; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: JS001 — JS001 240mg, i.v., q3w; Other name: Toripalimab
  Arms: JS001 Plus Nab-Paclitaxel
Drug: Nab-Paclitaxel — Nab-Paclitaxel 125 mg/m2, i.v., d1, d8, q3w
  Arms: JS001 Plus Nab-Paclitaxel
Drug: Placebo — Placebo, i.v., q3w;
  Arms: Placebo Plus Nab-Paclitaxel
Drug: Nab-Paclitaxel — Nab-Paclitaxel 125 mg/m2, i.v., d1, d8, q3w
  Arms: Placebo Plus Nab-Paclitaxel

SUMMARY:
This multicenter, randomized, double-blind study will evaluate the efficacy and safety of Toripalimab (JS001) combined with nab-paclitaxel compared with placebo combined with nab-paclitaxel for first/second line treatment of metastatic or recurrent triple-negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

Metastatic or recurrent triple negative breast cancer (TNBC);

* Histologically confirmed diagnosis of TNBC characterized by estrogen-receptor negative (ER-), progesterone receptor negative (PR-) and human epidermal growth factor-2 receptor negative (HER2-);
* Eligible for taxane monotherapy;
* No more than one line of chemotherapy in metastatic setting;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Life expectancy of 12 weeks or more;
* At least one measurable lesion per RECIST v1.1;
* Demonstrate adequate hematologic and organ functions as defined in the protocol

Exclusion Criteria:

Prior treatment with taxane as first line treatment;

* Prior treatment with PD-1 antibody, PD-L1 antibody, PD-L2 antibody, or CTLA4 antibody (or any other antibody acting on T cell co-stimulation or checkpoint pathway)
* MRI assessment during screening or previous imaging studies confirmed active or untreated brain metastases. Patients previously treated with local treatment of brain metastases has been stable for ≥ 1 month, and have stopped systemic hormonal therapy (>10 mg/d prednisone or equivalent) > 4 weeks before randomization can participate in the study;
* Meningeal carcinomatosis;
* Pregnancy or lactation;
* Active hepatitis B or hepatitis C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 531 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Intend to Treat patients. | Up to approximately 61 months from first patient in.
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the BIRC using RECIST v1.1, or death from any cause during the study, whichever occurs first. PD is defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 millimeter (mm) of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
PFS assessed by BICR using RECIST v1.1 in PD-L1 positive patients | Up to approximately 61 months from first patient in.
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death due to any cause during the study, whichever occurs first. PD is defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 millimeter (mm) of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) assessed by investigator using RECIST v1.1. Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | Up to approximately 61 months from first patient in.
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first. PD is defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 millimeter (mm) of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
Objective response rate (ORR) assessed by BICR or investigators using RECIST v1.1. Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | Up to approximately 61 months from first patient in.
  ORR is defined as the rate of CR(Complete Response) or PR (Partial Response), as determined by BICR using RECIST v1.1
Duration of response (DoR) assessed by BICR or investigators using RECIST v1.1. Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | Up to approximately 61 months from first patient in.
  DoR is defined as the time period from the date of initial CR or PR until the date of PD or death due to any cause, whichever occurs first.
Disease control rate (DCR) assessed by BICR or investigators using RECIST v1.1. Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | Up to approximately 61 months from first patient in.
  DCR is defined as the sum rate of CR, PR and SD (Stable Disease), as determined by BICR or investigators using RECIST v1.1
Overall Survival (OS). Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | Up to approximately 61 months from first patient in.
  OS is defined as the time from randomization to death from any cause
OS rate at 12 months. Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | Up to approximately 61 months from first patient in.
  OS is defined as the time from randomization to death from any cause.
OS rate at 24 months. Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | Up to approximately 61 months from first patient in.
  OS is defined as the time from randomization to death from any cause
Differences in safety and tolerability as assessed by the occurrence of adverse events. Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | From Day 1 to death from any cause, assessed up to end of study (up to approximately 46 months）
  From Day 1 to death from any cause, assessed up to end of study (up to approximately 61months）
Differences in the scores of disease/treatment-related symptoms evaluted by ECOG Performance Status. Analyzing among PD-L1 positive patients and Intend to Treat (ITT) respectively. | From Day 1 to death from any cause, assessed up to end of study (up to approximately 61months)
  Evaluated by Eastern Cooperative Oncogloy Group (ECOG) Performance Status

CONTACTS AND LOCATIONS:
Locations (53):
- China (53):
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Hebei University, Baoding
  - The first affiliated Hospital of Bengbu Medical College, Bengbu
  - Jilin Cancer Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Affiliated Hospital of Chengde Medical University, Chengde
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - The Second Hospital of Dalian Medical University, Dalian
  - The First People's Hospital of Foshan, Foshan
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Women and Children's Hospital of Guangdong Province, Guangzhou
  - The First Affiliated Hospital Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Province Hospital & The First Affiliated Hospital of USTC, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Second Hospital of Anhui Medical University, Hefei
  - Shandong Cancer Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Linyi Cancer Hospital, Linyi
  - The Affiliated Hospita of of Southwest Medical University, Luzhou
  - Jiangxi Cancer Hospital, Nanchang
  - The Third Hospital of Nanchang, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Changhai Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Liaoning Cancer Hospital&Intitute, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Cancer Hospital Affiliated to Xinjiang Medical University, Ürümqi
  - Hubei Cancer Hospital, Wuhan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Affiliated Hospital of Jiangnan University（Wuxi NO.4 People's Hospital）, Wuxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of The PLA Air Force Military Medical University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiangyang Central Hospital, Xiangyang
  - General Hospital of Ningxia Medical University, Yinchuan
  - Henan Provincial People's Hospital, Zheng'zhou
  - Henan Cancer Hospital, Zhengzhou